CLINICAL TRIAL: NCT03323905
Title: MRI-guided High Intensity Focused Ultrasound Ablation of Leiomyomas. Single Arm, Feasibility Study Using the Symphony - MRI Guided Focused Ultrasound System for the Treatment of Leiomyomas
Brief Title: Single Arm Study Using the Symphony -- MRI Guided Focused Ultrasound System for the Treatment of Leiomyomas
Acronym: HIFUSB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Sunnybrook Research Institute (Other); Arrayus Technologies Inc. (Industry)
Responsible Party: Principal Investigator, Dr. Elizabeth David, Affiliate scientist, Interventional Radiologist and Assistant Professor, Sunnybrook Health Sciences Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIFUSB
Record Dates: First submitted 2017-09-22; First posted 2017-10-27 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-07

CONDITIONS: Leiomyoma; Fibroid
MeSH Terms: conditions — Leiomyoma

STUDY DESIGN:
Intervention Model Description: Pilot single arm feasibility trial.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MR Guided High Intensity Focused Ultrasound (Experimental)
  Interventions: Device: Symphony MRI guided High Intensity Focused Ultrasound (HIFU)

INTERVENTIONS:
Device: Symphony MRI guided High Intensity Focused Ultrasound (HIFU) — The use of the MRI-HIFU for the ablation of leiomyomas

SUMMARY:
Single arm, first-in human feasibility study using the Symphony - MRI guided focused ultrasound system for the treatment of leiomyomas. The study is expected to accrue over 12 months. This study will help determine the feasibility to ablate leiomyomas, as measured by MR thermometry and contrast enhanced imaging. In addition, the study will look at the efficacy and safety of the treatment, as measured by the reduction in fibroid size and reduction in symptom severity score and adverse events. This study will help develop future pivotal trials using the same device.

ELIGIBILITY:
Inclusion Criteria:

1. MR-HFU device accessibility to fibroids that at least 50% of fibroid volume can be treated
2. Fibroids selected for treatment meet the following criteria

   1. Total planned ablation volume of all fibroids should not exceed 500 ml AND
   2. Completely non-enhancing fibroids should not be treated
3. Transformed SSS score >= 40
4. Pre- or peri-menopausal, as indicated by clinical evaluation
5. Weight < 140 kg or 310 lbs
6. Willing and able to attend all study visits
7. Willing and able to use reliable contraception methods
8. Uterine size < 24 weeks
9. Cervical cell assessment by PAP: normal, LOW Grade SIL, Low risk HPV or ASCUS subtypes of cervical tissue
10. Waist circumference <110cm or 43 inches

Exclusion Criteria:

1. Other Pelvic Disease (Other mass, endometriosis, ovarian tumor, acute pelvic disease, significant adenomyosis, prolonged bleeding requiring further evaluation as determined by patient's gynecologist)
2. Positive pregnancy test
3. Extensive scarring along anterior lower - abdominal wall (>50% of area)
4. Surgical clips in the potential path of the HIFU beam
5. Tattoos in the potential path of the HIFU beam
6. MRI contraindicated
7. MRI contrast agent contraindicated (including renal insufficiency)
8. Calcification around or throughout uterine tissue that may affect treatment
9. Communication barrier
10. Fibroids not quantifiable on MRI (e.g., multi-fibroid cases where volume measurements are not feasible)
11. Pedunculated fibroids
12. Bowel loops int he ultrasound beam path
13. Patients with inability to tolerate prolonged prone position for up to 3 hours
14. Patient with unstable medical conditions
15. Patients with coagulopathy or under current anti-coagulation therapy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 50 (Actual)
Dates: Start 2017-11-16 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-03-03 (Actual)

PRIMARY OUTCOMES:
The ability to ablate fibroid tissue measured by temperature elevation | 1 year
  Measured by MRI thermometry
The ability to ablate fibroid tissue indicated by Non-Perfused Volume (NPV) | 1 year
  Measure by contrast enhanced imaging
Safety of the system measured by collection of adverse events related to potential damage to tissue outside the treatment zone | 1 year
  Safety will be measured by collection of adverse events related to potential damage to tissue outside the treatment zone.
Safety of the system based on damage to skin measured by collection of adverse events related to potential damage to skin over the treatment volume | 1 year
  Safety will be measured by collection of adverse events related to potential damage to skin over the treatment volume.

SECONDARY OUTCOMES:
Treatment efficacy to reduce fibroid size | 1 year
  Reduction of fibroid volume in milliliters
Treatment efficacy to reduce fibroid size by NPV | 1 year
  Measured by non-perfused volume in milliliters
Treatment efficacy to reduce symptom severity by Symptom Severity Scores (SSS) | 1 year
  Change in symptoms to be quantified by Symptom Severity Scores (SSS) derived from Uterine Fibroid Symptom and Quality of Life questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: David Elizabeth, Principal Investigator — Sunnybrook Reserach Institute
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada